CLINICAL TRIAL: NCT01011166
Title: A Phase II, Randomized, Double-Blind Study to Evaluate the Safety and Antiviral Activity of IDX184 in Combination With Pegylated Interferon and Ribavirin in Subjects With Genotype 1 Chronic Hepatitis C Infection
Brief Title: Safety and Antiviral Activity of IDX184 in Combination With Pegylated Interferon and Ribavirin (MK-2355-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2355-004; IDX-08C-004 (Other: Idenix Protocol Number)
Record Dates: First submitted 2009-10-02; First posted 2009-11-11 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic Hepatitis C; HepC; Hep C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — IDX184; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- IDX184 50 mg QD + Peg-IFN/RBV (Experimental): Participants randomized 4:1 (active:placebo) to receive IDX184 50 mg or placebo once daily (QD) in combination with Peg-IFN/RBV on Days 14-28 and Peg-IFN/RBV on Days 14-28.
  Interventions: Drug: IDX184; Drug: Placebo; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)
- IDX184 100 mg QD + Peg-IFN/RBV (Experimental): Participants randomized 4:1 (active:placebo) to receive IDX184 50 mg or placebo QD in combination with Peg-IFN/RBV on Days 1-14 and Peg-IFN/RBV alone on Days 14-28.
  Interventions: Drug: IDX184; Drug: Placebo; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)
- IDX184 100 mg BID + Peg-IFN/RBV (Experimental): Participants randomized 4:1 (active:placebo) to receive IDX184 100 mg or placebo twice daily (BID) in combination with Peg-IFN/RBV on Days 1-14 and Peg-IFN/RBV alone on Days 14-28.
  Interventions: Drug: IDX184; Drug: Placebo; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)
- IDX184 150 mg QD + Peg-IFN/RBV (Experimental): Participants randomized 4:1 (active:placebo) to receive IDX184 150 mg or placebo QD in combination with Peg-IFN/RBV on Days 1-14 and Peg-IFN/RBV on Days 14-28.
  Interventions: Drug: IDX184; Drug: Placebo; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)
- IDX184 200 mg QD + Peg-IFN/RBV (Experimental): Participants randomized 4:1 (active:placebo) to receive IDX184 100 mg or placebo QD in combination with Peg-IFN/RBV on Days 1-14 and Peg-IFN/RBV on Days 14-28.
  Interventions: Drug: IDX184; Drug: Placebo; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)
- IDX184 200 mg BID + Peg-IFN/RBV (Experimental): Participants randomized 4:1 (active:placebo) to receive IDX184 200 mg or placebo BID in combination with Peg-IFN/RBV on Days 1-14 and Peg-IFN/RBV on Days 14-28.
  Interventions: Drug: IDX184; Drug: Placebo; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: IDX184 — IDX184 50 mg white opaque capsules taken by mouth from Day 1 to Day 14.
Drug: Placebo — Placebo white opaque capsules taken by mouth from Day 1 to Day 14.
Biological: Peginterferon alfa-2a (Peg-IFN) — Peg-IFN was supplied as 180 ug single-use, pre-filled syringes administered once weekly from Day 1 to Day 28.
  Other Names: Pegasys
Drug: Ribavirin (RBV) — RBV 200 mg capsules at a total daily dose of 1000 mg to 1200 mg (based on participant body weight) from Day 1 to Day 28.

SUMMARY:
This study will assess short term safety, antiviral activity and pharmacokinetics (PK) of IDX184 in combination with Peg-interferon (Peg-IFN)/Ribavirin (RBV) in participants with hepatitis C virus (HCV) genotype (GT) 1 infection. These data will guide dose selection for future, longer term studies.

ELIGIBILITY:
Inclusion Criteria:

* Has documented chronic HCV GT1 infection
* Agrees to use of double-barrier contraception and males agree not to donate sperm from the first dose of study therapy through at least 6 months after the final dose of study therapy

Exclusion Criteria:

* Has received previous antiviral treatment for HCV infection
* Has cirrhosis or decompensated liver disease
* Is pregnant or breastfeeding
* Is co-infected with hepatitis B virus (e.g., hepatitis B surface antigen [HBsAg] positive) and/or human immunodeficiency virus (HIV)
* Has clinically significant concomitant disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in HCV ribonucleic acid (RNA) level from Baseline to Day 15 | Baseline and Day 15
Percentage of participants experiencing adverse events (AEs) | Up to 28 days
Percentage of participants experiencing serious adverse events (SAEs) | Up to 28 days
Percentage of participants experiencing dose-limiting toxicities (DLTs) | Up to 28 days
Percentage of participants experiencing Grade 1-4 laboratory abnormalities | Up to 28 days

SECONDARY OUTCOMES:
Change in HCV RNA level from Baseline to Day 28 | Baseline and Day 28
Percentage of participants with undetectable HCV RNA at Day 15 | Day 15
Percentage of participants with undetectable HCV RNA at Day 28 | Day 28
Percentage of participants experiencing virologic breakthrough while on study therapy | Up to 28 days
Change in alanine aminotransferase (ALT) level from Baseline to Day 15 | Baseline and Day 15
Change in ALT level from Baseline to Day 28 | Baseline and Day 28
Maximum concentration (Cmax) | Up to 28 days
Time to maximum concentration (Tmax) | Up to 28 days
Area under the drug concentration-time curve (AUC) from time 0 to last measurable concentration (AUC0-t) | Up to 28 days
AUC from time zero to infinity (AUC0-~) | Up to 28 days
Trough concentration (Ctrough) | Up to 28 days
Observed terminal half-life (Thalf) | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lalezari J, Box T, O'Riordan W, Mehra P, Nguyen T, Poordad F, Dejesus E, Kwo P, Godofsky E, Lawrence S, Dubuc-Patrick G, Chen J, McCarville J, Pietropaolo K, Zhou XJ, Sullivan-Bolyai J, Mayers D. IDX184 in combination with pegylated interferon-alpha2a and ribavirin for 2 weeks in treatment-naive patients with chronic hepatitis C. Antivir Ther. 2013;18(6):755-64. doi: 10.3851/IMP2552. Epub 2013 Feb 25. PMID 23439365